CLINICAL TRIAL: NCT04191967
Title: Cervical Cancer Screening Among HIV-infected Women in Western Kenya: Evaluation of the Safety, Acceptability, and Efficacy of an Alternative Ablation Method for Treatment of Precancerous Lesions
Brief Title: Thermocoagulation for Treatment of Precancerous Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19405; 5D43TW009343 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Human Immunodeficiency Virus; HPV Infection; CIN 2/3
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Papillomavirus Infections | interventions — Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Thermocoagulation (Experimental): Thermal ablation of cervix for treatment of CIN2/3 among HIV-positive participants will be performed by a trained, non-physician clinician. Thermocoagulation will last approximately 20 seconds and will be performed using the Liger Thermocoagulator device
  Interventions: Device: Thermocoagulation

INTERVENTIONS:
Device: Thermocoagulation — Treatment of positive screening results will be performed using the Liger Thermocoagulator device
  Other Names: Liger thermocoagulator

SUMMARY:
The purpose of this study is to evaluate the safety, acceptability, and efficacy of Thermocoagulation for treatment of precancerous lesions among HIV-positive women in a screen-and-treat program in Western Kenya.

DETAILED DESCRIPTION:
Thermocoagulation is endorsed as an alternative to Cryotherapy for treatment of Visual Inspection with Acetic Acid (VIA) or Human Papillomavirus (HPV)-positive women by the 2018 Kenya national cancer guidelines.32 Data primary from Western countries demonstrate similar efficacy for the treatment of precancerous lesions between Cryotherapy and Thermocoagulation. Data on safety, acceptability, and efficacy, particularly linked to gold-standard pathology, among HIV-positive women in low-resource settings are scare. Given the demonstrated benefits over cryotherapy including increased portability and availability hence easier implementation, use of thermal coagulation for the treatment of precancerous lesions in low resource settings could significantly improve access to treatment compared with cryotherapy.

This study seeks to fill a critical data gap by evaluating the efficacy of thermocoagulation among HIV-positive positive women using gold-standard biopsy for disease verification at baseline and follow-up, as indicated. We will also assess the safety and acceptability of this treatment modality among patients and providers

Aim 1: To evaluate the efficacy of thermal coagulation for the treatment of HIV-positive, HPV-positive women by assessing rates of HPV persistence and CIN2/3 rate at 12 months after treatment

Aim 2: To evaluate the safety and acceptability of thermal coagulation for treatment of abnormal cervical lesions within a screen-and-treat program among HIV-positive women in Western Kenya.

Aim 3: Evaluate provider acceptability of thermal coagulation for the treatment of precancerous cervical lesion within a screen-and-treat program in Western Kenya.

Outline:

Counseling on HPV, cervical cancer, and the screening process was offered during routine HIV clinics in group and individual settings. Participants will then be provided self-sampling instructions, a collection kit, and a private area to perform self-collection. The self-collected HPV samples will be labeled, stored, and processed for DNA of 14 high-risk HPV types. HPV-positive participants were invited for a return visit, including a pelvic examination and visual inspection with acetic acid (VIA) to determine eligibility for ablative therapy. After ablation, a questionnaire will be administered to participants to evaluate treatment experience. All participants will be given a 4- to 6-week phone or in-person follow-up appointment, per participant preference

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-65 years.
2. Enrolled in HIV care at FACES-supported clinics in Kisumu County.
3. Able to understand a written informed consent document, and willing to sign it.
4. Speaks a language that the consent form and data collection instruments are written in.

Exclusion Criteria:

1. Has a history of cervical cancer.
2. Has received any treatment for cervical precancer after screening positive for precancer.
3. Has evidence of cervical infection.
4. Pregnant women are excluded from this study.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chemtai Mungo, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mungo C, Osongo CO, Ambaka J, Randa MA, Omoto J, Cohen CR, Huchko M. Safety and Acceptability of Thermal Ablation for Treatment of Human Papillomavirus Among Women Living With HIV in Western Kenya. JCO Glob Oncol. 2020 Jul;6:1024-1033. doi: 10.1200/GO.20.00035. PMID 32634066
- [Derived] 2022 ASCCP Poster Presentations. J Low Genit Tract Dis. 2022 Apr 1;26(2S):6-13. doi: 10.1097/LGT.0000000000000671. No abstract available. PMID 35350043
- [Derived] Mungo C, Osongo CO, Ambaka J, Randa MA, Samba B, Ochieng CA, Barker E, Guliam A, Omoto J, Cohen CR. Feasibility and Acceptability of Smartphone-Based Cervical Cancer Screening Among HIV-Positive Women in Western Kenya. JCO Glob Oncol. 2021 May;7:686-693. doi: 10.1200/GO.21.00013. PMID 33999653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2019 and February 2020, women enrolled in care at Fostering Advances through Collaboration, Education & Sciences (FACES)- supported HIV clinics in western Kenya were recruited to the study.
Pre-assignment Details: All participants received cervical cancer screening using human papillomavirus (HPV) testing. Participants with positive results received a biopsy and then proceeded to same-day treatment. Thermocoagulation candidates must have a fully visualized, squamocolumnar junction, cervical lesions (if present) covering < 75% of cervix, and no endocervical component of lesion, or suspicion for cancer. Participants who were not candidates for ablation were referred to a nearby facility.
Period: Screening & Thermocoagulation (Ablation)
Arm/Group | Thermocoagulation
Started | 379 (Participants screened for cervical cancer using HPV testing)
Completed | 293
Not Completed | 86
Not completed — Not considered candidates for thermocoagulation | 86
Period: 12 Month Follow-up
Arm/Group | Thermocoagulation
Started | 58
Completed | 54
Not Completed | 4
Not completed — Pathology results for 12 month treatment efficacy not available for these participants | 4

BASELINE CHARACTERISTICS:
Population: Candidates for ablation must had had a fully visualized, squamocolumnar junction; cervical lesions, if present, that covered < 75% of the cervix; and no endocervical component of the lesion or suspicion for cancer.
Arm/Group | Thermocoagulation
Number analyzed (Participants) | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 293
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 293
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 293
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Kenya | 293
Prior cervical cancer screening [Number; unit: participants] | 206

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With no Evidence of Cervical Dysplasia at 12-months
Description: The proportion of participants with no evidence of cervical dysplasia at 12-months follow-up, defined as biopsy-conﬁrmed CIN1 result or normal ﬁndings, 12-months following treatment.
Time Frame: 12 months
Measure: Number; unit: proportion of participants
Groups:
- Thermocoagulation: Thermal ablation of cervix for treatment of CIN2/3 among HIV-positive participants will be performed by a trained, non-physician clinician.Thermocoagulation will last approximately 20 seconds and will be performed using the Liger Thermocoagulator device
Arm/Group | Thermocoagulation
Number analyzed (Participants) | 54
proportion of participants | 0.66

2. Primary Outcome: Proportion of Participants With Persistent HPV at 12-month Follow-up
Description: The proportion of persistence of HPV at follow-up will be reported defined as treatment failure with persistent biopsy-confirmed CIN2/3.
Time Frame: 12 months
Measure: Number; unit: proportion of participants
Arm/Group | Thermocoagulation
Number analyzed (Participants) | 54
proportion of participants | 0.34

3. Secondary Outcome: Frequency of Pain Score Category
Description: A 4-point Visual Analog Scale (VAS) for pain assessment was used to evaluate pain immediately after treatment. The pain VAS was comprised of verbal descriptors, one for each symptom extreme. The pain VAS is self-completed by the respondent. The respondent is asked to select the point that represents their pain intensity. The "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. The following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
Time Frame: Day of Treatment, approximately 1 day
Measure: Count of Participants; unit: Participants
Groups:
- Thermocoagulation: Thermal ablation of cervix for treatment of CIN2/3 among HIV-positive women
  Thermocoagulation: Treatment of positive screening results will be performed using the Liger Thermocoagulator device
Arm/Group | Thermocoagulation
Number analyzed (Participants) | 293
Participants
  No pain | 15
  Mild pain | 231
  Moderate pain | 42
  Severe pain | 5

4. Secondary Outcome: Percentage of Participants Reporting Treatment-related Adverse Events (AE)
Description: The percentage of participants reporting grade 2 and higher AEs, and severe adverse events (SAEs) during the 4-week follow-up will be reported by event.
Time Frame: Up to 6 weeks following treatment
Measure: Number; unit: percentage of participants
Arm/Group | Thermocoagulation
Number analyzed (Participants) | 293
percentage of participants
  Bleeding | 4
  Vaginal Discharge | 51.2
  Pelvic Pain | 19.6
  Participants with Grade 3 or 4 adverse events | 0

5. Secondary Outcome: Frequency of Positive Participant Satisfaction Responses
Description: Participant satisfaction with thermocoagulation will be evaluated by determining the proportion of participants indicating a response of 'yes' to the question "Do you feel satisfied with the treatment you received?" with an alternative response of 'no' at the 4-6 week follow-up visit.
Time Frame: Up to 6 weeks following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Thermocoagulation
Number analyzed (Participants) | 293
Participants | 292

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Adverse events (AEs) were graded using the Division of AIDS, National Institute of Allergy and Infectious Diseases: Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events: Corrected version 2.1. (https://rsc.niaid.nih.gov/sites/default/files/daidsgradingcorrectedv21.pdf).
Arm/Group | Thermocoagulation
All-Cause Mortality (participants affected / at risk) | 0/293
Serious Adverse Events (participants affected / at risk) | 0/293
Other Adverse Events (participants affected / at risk) | 262/293
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Thermocoagulation (N=293)
Vaginal hemorrhage (Reproductive system and breast disorders) | 99
Vaginal discharge (Reproductive system and breast disorders) | 258
Pain (not associated with study agent injections-not specified elsewhere (Injury, poisoning and procedural complications) | 1 — Backache
Pelvic Pain (Reproductive system and breast disorders) | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/67/NCT04191967/Prot_SAP_001.pdf
  • Informed Consent Form (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04191967/ICF_000.pdf